CLINICAL TRIAL: NCT00005492
Title: Pooled Analysis of NHANES I/II--Race, Gender, and CHD
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5009; R03HL058436 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

SUMMARY:
To conduct a pooled analysis of NHANES I/II data on race, gender, and coronary heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

Over the last 25 years, a sustained and marked decline in death rates from coronary heart disease (CHD) has occurred for all major segments of the U.S. population. Recently, however, the decline has proceeded less rapidly in blacks than in whites, and in women than men. These trends have focused further attention on possible heterogeneity in the risk factor patterns among the demographic sub-groups. Previous studies of CHD risk factors in blacks and whites using the First National Health and Examination Survey Epidemiologic Follow-up Study (NHEFS-I, 11-year follow-up), including this group's own work, demonstrate its potential strengths, while at the same time foundering on the problem of low statistical power. With the extension of the follow-up of NHANES-I cohort (1971-1974) to 1987 (14 years) and the completion of 14-year follow-up for NHANES II cohort (1976-1980), a strong rationale exists to undertake a "pooling project." The resulting data set would provide optimal characterization of CHD risk at the national level.

DESIGN NARRATIVE:

The study sought to determine whether data from NHANES I and NHANES II could be pooled. To accomplish this, the distribution of baseline measures was assessed and a determination was made whether the same logistic prediction equations fitted both studies. Also, gender-race differences were examined in individual exposure-outcome relationships, patterns of co-morbidity, and population attributable risks.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-08; Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Youlian Liao — Loyola University

REFERENCES:
- [Background] Liao Y, McGee DL, Cooper RS, Sutkowski MB. How generalizable are coronary risk prediction models? Comparison of Framingham and two national cohorts. Am Heart J. 1999 May;137(5):837-45. doi: 10.1016/s0002-8703(99)70407-2. PMID 10220632